CLINICAL TRIAL: NCT00429169
Title: Paroxetine Versus Bupropion for Suicide Ideators or Attempters With Major Depressive Disorder
Brief Title: Paroxetine/Bupropion in Suicide Attempters/Ideators With Major Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed differential treatment effects.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Grunebaum, MD, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5933R; K23MH076049 (NIH); DSIR 8KRT-AT
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Depression
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Paroxetine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine (Active Comparator): Participants will receive paroxetine for 8 weeks
  Interventions: Drug: Paroxetine
- Bupropion (Active Comparator): Participants will receive bupropion for 8 weeks
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Paroxetine — Dosage will be 25 mg every day for 2 weeks, then 37.5 mg every day for 2 weeks, and then optional increase to 50 mg every day for the remainder of treatment.
  Other Names: Paxil CR
  Arms: Paroxetine
Drug: Bupropion — Dosage will be 150 mg every day for 2 weeks, then 300 mg every day for 2 weeks, and then optional increase to 450 mg every day for the remainder of treatment.
  Other Names: Wellbutrin XL
  Arms: Bupropion

SUMMARY:
The primary study comparing effectiveness for suicidal ideation and/or behavior of two antidepressant medications in depressed patients who have attempted suicide or are currently experiencing suicidal thoughts has been completed.

A secondary study component using functional magnetic resonance imaging (fMRI) to investigate different medication effects on reward processing in the same sample is ongoing.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common and serious psychiatric illness. It is among the leading causes of disability and is the psychiatric disorder most often associated with suicide. The treatment of MDD with antidepressant medication remains largely trial and error. Little empirical evidence exists to guide the treatment of MDD when suicide risk is a major factor. Selective serotonin reuptake inhibitors (SSRIs) are a type of antidepressant medication that works by increasing the amount of serotonin, a natural substance in the brain that helps maintain mental balance. The study compared the effectiveness of paroxetine, an SSRI, versus bupropion, a non-SSRI, on suicidal ideation and/or behavior in depressed patients with a past suicide attempt and/or current suicidal thoughts. Results of the completed primary study have been published (Grunebaum MF et al. Neuropsychopharmacology. 2012 Feb;37(3):697-706).

In the ongoing secondary neuro-imaging component of the study, Participants are randomly assigned to either paroxetine or bupropion treatment for 8 weeks with fMRI scans involving a reward processing task at baseline and Week 8. Weekly study visits include interviews with a psychologist, self-report scales, and medication monitoring. All participants will then be offered 4 additional months of open clinical treatment. If original medication assignments prove to be ineffective, participants will have the option to switch to another medication. After completing the study, participants will be referred for ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from a major depressive episode (unipolar only)
* History of a past suicide attempt or score greater than 2 on the Hamilton Depression Rating Scale (HDRS) item #3 (suicide) at in-person screening interview. Patients with suicidal plan or intent will only be enrolled as inpatients if independent inpatient treatment team agrees.
* Patients 60 years of age and older must score at least 25 on MMSE at screening.
* Patients 60 years of age and older must have a normal ECG within the past year.

Exclusion Criteria:

* Any of the following conditions: bipolar disorder; current psychotic symptoms; bulimia or anorexia that is current or within the past year, or current purging at least twice a week for three months; already taking selective serotonin reuptake inhibitors (SSRIs) or bupropion for other indications (such as anxiety disorders)
* Primary disorder is an anxiety disorder (e.g., panic disorder, general anxiety disorder, obsessive compulsive disorder, social anxiety disorder), with secondary depression
* Drug or alcohol dependence within 6 months prior to study entry (current drug or alcohol abuse may be permitted if study officials determine that the abuse is of lesser importance than the major depressive episode)
* Systolic blood pressure greater than or equal to 140 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg
* Significant active physical illness, particularly those that may affect the brain or serotonergic system (e.g., blood dyscrasias lymphomas, hypersplenism, endocrinopathies, kidney failure, severe chronic obstructive lung disease, autonomic neuropathies, active malignancy)
* Active medical problems
* Requires antipsychotic medication
* History of hypomania or mania while taking antidepressants
* Any condition that may make the use of an SSRI or bupropion medically inadvisable
* Currently using Zyban
* Failure to respond to adequate trials of three SSRIs, paroxetine, or bupropion within 2 years prior to study entry (failure to respond to therapeutic trial defined as at least 2/3 maximal daily dose [PDR] for at least 6 weeks)
* Pregnant, breastfeeding, or plans to become pregnant during the course of study participation
* Currently on effective treatment, requires adjunctive antipsychotic or mood stabilizing medication, or is unlikely to respond to single agent treatment for depression
* Patients with ferrous metal implants in their bodies, or a history of claustrophobia that precludes MRI, will be excluded.
* Patients assessed as being unlikely to tolerate the maximum 2-week delay to start of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2004-06; Primary Completion 2010-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Grunebaum, MD, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Grunebaum MF, Ellis SP, Duan N, Burke AK, Oquendo MA, John Mann J. Pilot randomized clinical trial of an SSRI vs bupropion: effects on suicidal behavior, ideation, and mood in major depression. Neuropsychopharmacology. 2012 Feb;37(3):697-706. doi: 10.1038/npp.2011.247. Epub 2011 Oct 12. PMID 21993207
- [Derived] Grunebaum MF, Keilp JG, Ellis SP, Sudol K, Bauer N, Burke AK, Oquendo MA, Mann JJ. SSRI versus bupropion effects on symptom clusters in suicidal depression: post hoc analysis of a randomized clinical trial. J Clin Psychiatry. 2013 Sep;74(9):872-9. doi: 10.4088/JCP.12m08000. PMID 24107760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates were 2/2005-7/2009 with follow-up completed in January 2010.
Pre-assignment Details: N=101 subjects enrolled, but N=23 did not return after enrollment, so N=78 were randomized.
Period: Overall Study
Arm/Group | Paroxetine | Bupropion
Started | 38 | 40
Completed | 36 (2 subjects excluded due to re-diagnosis/ineligibility.) | 38 (2 subjects excluded: re-diagnosis/ineligibility (1), and did not return after randomization (1).)
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Ineligibility discovered after entry | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine | Bupropion | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 38 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.8) | 37.9 (11.9) | 36.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Go-No go Test
Description: Change in neuropsychological measure of impulsivity. Computer-based task involving induction of a dominant response tendency and testing of the subject's ability to withhold responding to less frequent non-target stimuli.
Time Frame: Measured at Baseline and Week 8
Population: These were the number with analyzable data
Measure: Mean (Standard Deviation); unit: Commission errors
Arm/Group | Paroxetine | Bupropion
Number analyzed (Participants) | 30 | 27
Commission errors | -0.09 (0.8) | -0.06 (0.89)

2. Primary Outcome: Scale for Suicidal Ideation
Description: The clinician-rated Beck Scale for Suicidal Ideation (SSI) (Beck et al 1979)was used weekly for 8 weeks. It has 19 items scaled 0 (least severe) to 2 (most severe) and total score is the sum, ranging 0 to 38 (Beck et al 1979). Items measure frequency, intensity, and attitudes toward suicidal thoughts, feelings of control over them, and suicide plans. Mean score in 90 inpatients hospitalized for suicidal ideation was 9.4±8.4, versus 4.4±5.8 in outpatients as cited in the study by Beck et al, 1979.
Time Frame: Baseline and Week 8
Population: The study was powered for N=50 subjects per group based on naturalistic pilot data from our clinic. An interim data analysis showed an interaction of treatment with baseline suicidal ideation severity on follow-up ideation. After consulting with clinical colleagues, statisticians and the IRB, a decision was made to stop enrollment.
Measure: Mean (Standard Deviation); unit: Points on Scale for Suicidal Ideation
Groups:
- Paroxetine: Paroxetine acute treatment for 8 weeks.
- Bupropion: Bupropion acute treatment for 8 weeks.
Arm/Group | Paroxetine | Bupropion
Number analyzed (Participants) | 36 | 38
Points on Scale for Suicidal Ideation
  Baseline | 8.0 (6.7) [-0.57 to -0.023] | 9.9 (7.4)
  Week 8 | 2.3 (4.5) | 4.7 (6.6)
Statistical Analysis 1: Comparison: Paroxetine vs Bupropion; Generalized least squares model of Scale for Suicidal Ideation score during 8-week acute treatment of major depressive disorder; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — The p-value applies to the interaction term of Treatment X Baseline Suicidal Ideation severity; regression coefficient = -0.29, 95% CI 2-sided [-0.57 to -0.023]

3. Primary Outcome: Occurrence of Suicidal Ideation or Acts Necessitating a Change in Treatment
Description: Suicide attempts, other suicidal behavior, or increase in suicidal thoughts that required a change in clinical treatment.
Time Frame: Measured at Month 6
Population: These were the number of subjects with analyzable data.
Measure: Number; unit: Events
Arm/Group | Paroxetine | Bupropion
Number analyzed (Participants) | 36 | 38
Events | 4 | 6

4. Primary Outcome: Brain Activity Measured by BOLD Signal With fMRI During a Reward Processing Task.
Description: Comparison of fMRI results at baseline and after 8 weeks of antidepressant pharmacotherapy with paroxetine vs. bupropion.
  Percent change in contrast of parameter estimates (COPE). COPE is measured during Monetary Incentive Delay Task.
  Task conditions are:
  Reward=BOLD signal when subject wins 5 cents vs. wins 0 cents Punishment=BOLD signal when subject loses 5 cents vs. loses 0 cents
Time Frame: Baseline and Week 8.
Population: Major depressive disorder with suicidal thoughts or past suicide attempt.
Measure: Mean (Full Range); unit: percentage of change in COPE
Arm/Group | Paroxetine | Bupropion
Number analyzed (Participants) | 4 | 3
percentage of change in COPE | -0.27 [-0.59 to 2.9] | -0.95 [-1.3 to 1.7]

ADVERSE EVENTS:
Arm/Group | Paroxetine | Bupropion
Serious Adverse Events (participants affected / at risk) | 3/36 | 2/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine (N=36) | Bupropion (N=38)
Suicide attempt by acetaminophen overdose (Hepatobiliary disorders) | 1 (1) | 0 (0) — Patient admitted to hospital and treated. No serious medical sequelae resulted.
Increased suicidal thoughts causing admission to hospital (Nervous system disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
1. Significant dropout meant the number of subjects with analyzable data was smaller than the number enrolled.
2. An interim analysis of this pilot study showed differential treatment effects so a decision was made to stop enrollment early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No